CLINICAL TRIAL: NCT04903665
Title: Gynecologic Malignancies Early-stage Detection by Liquid Biopsy in Peripheral Blood: a Prospective, Observational Study
Brief Title: PERformance of Multi-Cancer Early-detectIon Based on Various Biomarkers in fEmale Cancers, PERCEIVE-I
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Collaborators: Guangzhou Burning Rock Bioengineering Ltd. (Industry)
Responsible Party: Principal Investigator, Xiaohua Wu MD, Director, Fudan University
Other Study IDs: FDZL-2021002
Record Dates: First submitted 2021-05-24; First posted 2021-05-26 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Gynecologic Cancer
Keywords: gynecologic cancer; early detection; liquid biopsy; cell-free DNA

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, white blood cells and formalin fixed, paraffin embedded (FFPE) tumor tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer Arm: Participants with new diagnosis of gynecologic cancers, from whom blood samples will be collected.
  Interventions: Device: Multi-cancer early detection test
- Benign Arm: Participants with new diagnosis of benign gynecologic diseases, from whom blood samples will be collected.
  Interventions: Device: Multi-cancer early detection test

INTERVENTIONS:
Device: Multi-cancer early detection test — Blood collection and multi-cancer early detection testing

SUMMARY:
This study is a prospective study aimed to develop and validate the performance of combined multi-omitcs assays for early detection of gynecologic cancers. Biomarkers of cfDNA methylation, ctDNA mutation and blood miRNA markers will be evaluated. The study will enroll approximately 495 female participants, including participants with gynecologic cancers or benign diseases.

ELIGIBILITY:
Inclusion Criteria for Cancer Arm Participants:

* Age 18 years or older
* Able to provide a written informed consent
* Confirmed diagnosis or highly suspicious cases of gynecologic malignancies
* No prior or ongoing anti-cancer therapy (local or systematic) prior to study blood draw

Exclusion Criteria for Cancer Arm Participants:

* Pregnancy or lactating women
* Recipients of organ transplant or prior non-autologous (allogeneic) bone marrow transplant or stem cell transplant
* Recipients of blood transfusion within 7 days prior to study blood draw
* Recipients of any anti-cancer therapy within 30 days prior to study blood draw, due to diseases other than cancer

Inclusion Criteria for Benign Arm Participants:

* Age 18 years or older
* Able to provide a written informed consent
* Confirmed diagnosis of benign gynecologic diseases
* No prior radical treatment of the benign diseases prior to study blood draw

Exclusion Criteria for Benign Arm Participants:

* Pregnancy or lactating women
* Recipients of organ transplant or prior non-autologous (allogeneic) bone marrow transplant or stem cell transplant
* Recipients of blood transfusion within 7 days prior to study blood draw
* Recipients of any anti-cancer therapy within 30 days prior to study blood draw, due to diseases other than cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants will be recruited from the participating medical center and assigned into two arms, including participants with new diagnosis of gynecologic malignancies and benign gynecologic diseases.
Sampling Method: Non-Probability Sample
Enrollment: 495 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2022-08-22 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity,specificity and tissue of origin accuracy of the multi-omics model as early detection for gynecologic cancers. | 12 months

SECONDARY OUTCOMES:
Sensitivity and specificity of the multi-omics model in early detection of gynecologic cancers in different stages. | 12 months
Sensitivity and specificity of the multi-omics model in early detection of different gynecologic cancer diseases | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Wu, M.D.&Ph.D, Principal Investigator — Department of Gynecological Oncology, Fudan University Shanghai Cancer Center
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China